CLINICAL TRIAL: NCT01496560
Title: Comparison of Procedural Sequence in Same Day Consecutive Bidirectional Endoscopy Using Moderate Sedation: A Prospective Randomized Study
Brief Title: Open Prospective Study for Determination of Predictive Measures for Pain During Colonoscopy
Status: Withdrawn | Type: Observational
Why Stopped: study terminated due toTechnical issue pre -recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Dan Carter, Gastroenterologist, Gastroenterologist, Sheba Medical Center
Other Study IDs: Sheba-11-8679-DC-CTIL
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Pain
Keywords: colonoscopy; pain; rectal balloon
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to determine what precolonoscopic measures can be correlated to pain during colonoscopy

DETAILED DESCRIPTION:
The aim of the work is to determine prdictive pre-endoscopic factors for pain during colonoscpy. These factors may be demographic, antrophometric, socio-ecomomic, related to previous medical staus or to anxiety levels.

We will try to find an objective parameter for prdiction of pain during colonoscopy, so pre-procedural intervantion will be applied in order to reduce the pain.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70
* screening colonoscopy

Exclusion Criteria:

* Failed prior colonoscopy
* pain as a main referral indication
* complications during previous exam
* Inpatients
* Excision of more than 3 polyps
* Diagnosis ofCancer, IBD
* Incomplete exam

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing screening colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pre-endoscopic Rectal balloon volumes | 1 year
  Volume for first sensation, desire to deficate and maximal tolerance volume

SECONDARY OUTCOMES:
Demographic data | 1 year
  Demographic data related to excessive pain
Pre-endocopic levels of anxiety | 1 year
  Relation of Pre-endoscopic levels of anxiety to pain during colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Dan Carter, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel

REFERENCES:
- [Background] Park DI, Kim HJ, Park JH, Cho YK, Sohn CI, Jeon WK, Kim BI, Ryu SH, Sung IK. Factors affecting abdominal pain during colonoscopy. Eur J Gastroenterol Hepatol. 2007 Aug;19(8):695-9. doi: 10.1097/01.meg.0000219097.32811.24. PMID 17625440